CLINICAL TRIAL: NCT04260074
Title: Biomarkers in Head and Neck Cancer - Epigenetic Changes and Hypermethylation of Promoter-regions
Brief Title: Epigenetic Changes in Head and Neck Cancer
Status: Completed | Type: Observational
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Christian Sander Danstrup, Associate Professor, M.D., Aalborg University Hospital
Other Study IDs: N-20190047
Record Dates: First submitted 2020-02-05; First posted 2020-02-07 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Head and Neck Cancer; Squamous Cell Carcinoma; Head and Neck Squamous Cell Carcinoma; Head and Neck Neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Squamous Cell; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biopsies from tumour and healthy buccal mucosa. Blood samples from both case and control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Oral Cancer group: 20 consecutive patients with oral squamous cell carcinoma referred to the Department of Otolaryngology - Head and Neck Surgery
- Healthy oral mucosa group: 20 controls with normal buccal mucosa upon examination.

SUMMARY:
With this study, the investigators will investigate the epigenetic changes, which may contribute to the development of head and neck squamous cell carcinomas.

ELIGIBILITY:
Cancer group:

Inclusion Criteria :

* Written informed consent
* Histologically confirmed oral squamous cell carcinoma

Exclusion Criteria:

* History of cancer
* Uncontrolled comorbidity

Control group:

Inclusion Criteria :

* Written informed consent
* Normal buccal mucosal surface.
* Normal ENT-examination

Exclusion Criteria:

* History of cancer
* Uncontrolled comorbidity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cancergroup:
  Patients referred to The Department of Otolaryngology - Head and Neck surgery
  Controlgroup:
  Patients referred to a private clinic for oral and maxillofacial surgery
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2021-07-14 (Actual); Study Completion 2021-07-14 (Actual)

PRIMARY OUTCOMES:
Differences in epigenetic changes | 6 months
  Differences between tumor- and healthy group

CONTACTS AND LOCATIONS:
Overall Officials: Michael Gaihede, Professor, Principal Investigator — Department of Otolaryngology - Head and Neck Surgery
Locations (1):
- Department of Otolaryngology - Head and Neck Surgery, Aalborg, Denmark